CLINICAL TRIAL: NCT03721042
Title: Demonstrating the Diagnostic Power of an Electronic Nose: Pilot Study on Exhaled Air Samples
Brief Title: Demonstrating the Diagnostic Power of an Electronic Nose: Study on Exhaled Air Samples
Acronym: OLFADIAG
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: no PI to continue the study
Sponsor: Nouvelle Clinique Bonnefon (Other)
Collaborators: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: HSM_NCB_2018-1; NCT03715855 (obsolete NCT alias)
Record Dates: First submitted 2018-10-25; First posted 2018-10-26 (Actual); Last update posted 2022-04-14 (Actual); Status verified 2022-04

CONDITIONS: Alzheimer Disease; Gastric Cancer; Urologic Cancer; Pneumological Cancer
MeSH Terms: conditions — Alzheimer Disease; Stomach Neoplasms; Urologic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- exhaled air (Experimental): exhaled air analysis of patients
  Interventions: Device: olfactory measuring device

INTERVENTIONS:
Device: olfactory measuring device — Patients blowing into bags then analysis by olfadiag system

SUMMARY:
The investigators don't know yet how the nose and the brain decode the smells. Scientific studies in neuroscience have shown that people who have tumors may have changes in the smell of secretions. Dogs are extremely efficient at detecting these changes, even before imaging studies. A review of the recent literature shows the different work done on the diagnosis of dogs on human pathologies, especially oncology. It is now known that the smell of exhaled gases is representative of the intestinal biotope and that a large number of pathologies are related to the type of microbial populations that inhabit the intestines.

Copying the olfactory organs could thus be of major interest for the early diagnosis of pathologies. More and more works are interested in the diagnostic power of electronic noses. From a technical point of view, these are nano-sensors that mimic the olfactory receptors from the breath gas of the subjects. They analyze the molecules present and compare them with a database to establish a diagnosis according to a probabilistic algorithm.

The use of exhaled air for the diagnosis of cancerous pathologies has already been the subject of scientific work. A classification using the SVM (support vector machine) method using data from 320 sensors made it possible to differentiate patients with lung cancer from controls in 98.8% of cases. The differential diagnosis of obstructive bronchopneumopathy was also very well done in this same study. Another study shows equally encouraging results, highlighting sensitivities and specificities above 80%.

ELIGIBILITY:
Inclusion Criteria:

* The patient must have signed the free and informed consent form or their guardian if applicable. If the state of health of the patient does not allow him to give and sign his consent, it will be sought from the person of trust
* The patient must be an affiliate or beneficiary of a health insurance plan
* The patient is at least 18 years old

Exclusion Criteria:

* The patient participates or has participated within 3 months in another study that may have modified their intestinal biotope
* The patient is in an exclusion period determined by a previous study
* The patient is under the protection of justice
* The patient or guardian or trusted person refuses to sign the consent
* The patient does not read the French language fluently
* The patient claims to be pregnant
* The patient is breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2018-10-11 (Actual); Primary Completion 2019-11-05 (Actual); Study Completion 2020-10-01 (Actual)

PRIMARY OUTCOMES:
positive predictive value and negative predictive value | 18 months
  positive predictive value and negative predictive value of the electronic nose

CONTACTS AND LOCATIONS:
Locations (1):
- Nouvelle Clinique Bonnefon, Alès, France

IPD SHARING:
Plan to Share IPD: No